CLINICAL TRIAL: NCT01409382
Title: Repercussion of Maternal Lifestyle on Obstetric and Neonatal Outcomes
Brief Title: Maternal Lifestyle and Neonatal Hypoglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital dos Servidores do Estado do Rio de Janeiro (Other Government)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Silvia Hoirisch Clapauch, Principal investigator, Hospital dos Servidores do Estado do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 000416-09-08-2010
Record Dates: First submitted 2011-05-27; First posted 2011-08-04 (Estimated); Results first posted 2016-01-21 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-08

CONDITIONS: Hyperinsulinemia; Miscarriages; Pregnancy; Sedentary Lifestyle; Hypoglycemia
Keywords: neonatal hypoglycemia; pregnancy; physical activity; sedentary lifestyle; high-glycemic index diet; take-home baby; recurrent miscarriages; preterm delivery
MeSH Terms: conditions — Hyperinsulinism; Abortion, Spontaneous; Sedentary Behavior; Hypoglycemia; Motor Activity; Abortion, Habitual; Premature Birth

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Active Comparator): Daily brisk walking plus a carbohydrate-restricted diet
  Interventions: Behavioral: Daily brisk walking plus a carbohydrate-restricted diet
- Standard follow-up (No Intervention): Prenatal care will proceed according to the routine.

INTERVENTIONS:
Behavioral: Daily brisk walking plus a carbohydrate-restricted diet — Daily brisk walking at moderate speed (4 km/h) for at least 40 minutes per day, 7 days a week. Patients will be recommended to avoid high-glycemic index meals (such as snacks, candies, fiber-free juices and sugar-sweetened beverages), and to eat at least two daily servings of meat, poultry, fish (e.g. 2 g/kg) or other protein-rich food, starting when they decided to get pregnant and continuing until delivery. Recommendations will be emphasised at every appointment. Antidepressants will not be discontinued in both groups, but patients on paroxetine and sertraline, will be switched to fluoxetine.
  Arms: Lifestyle counseling

SUMMARY:
tPA has a pivotal role in placentation, mediationg activation of growth factors, such as vascular endothelial growth factor and brain-derived neurotrophic factor, degradation of extracellular matrix and basement membrane (directly or through activation of matrix metalloproteinases) and formation of hemidesmosomes.

A high-carbohydrate intake combined with lack of physical activity provides a strong stimulus for maternal insulin production. In this scenario, either β-cells are dysfunctional and diabetes supervenes, or excessive amounts of insulin are produced, providing pathological stimulation of PAI-1 synthesis. Given that PAI-1 is a major tPA inhibitor, PAI-1 excess may affect placentation, increasing the risk of first trimester losses, preterm deliveries and intrauterine growth restriction.

Our hypothesis was that prematurity was not the cause of neonatal hypoglycemia, but a parallel occurrence of a strong stimulus for maternal, fetal and neonatal production of insulin.

DETAILED DESCRIPTION:
In an observational study, we sought to determine whether markers of hyperinsulinemia or situations that increase maternal insulin requirements would increase the risk of neonatal hypoglycemia. Mothers were selected if they had grade III obesity, acanthosis nigricans (surrogates of chronic maternal hyperinsulinemia), any invasive bacterial infection or if they had used corticosteroid within seven days before delivery (surrogates of subacute insulin resistance), if they reported to have consumed a high-glycemic index diet within 24 hours before delivery or if they were physically inactive within 24 hours before delivery (conditions that could increase maternal insulin requirements close to delivery).

Based on the finding that that the risk of neonatal hypoglycemia increased fivefold with inactivity (95% CI: 2-11, P <0.001), 11-fold with high-carbohydrate intake (95% CI: 4-24, P <0.001) and 329-fold with both risk factors (95% CI: 32-3362, P <0.001), next we have evaluated how a protocol combining exercises and a balanced diet throughout pregnancy influences maternal and neonatal outcomes. One of the outcomes analyzed was neonatal hypoglycemia.

ELIGIBILITY:
Inclusion criteria: recurrent early unexplained miscarriages Exclusion criteria: (i) antiphospholipid antibodies, (ii) second- or third-trimester losses, (iii) multiple pregnancy, (iv) anatomical abnormalities that could increase the risk of early miscarriages, (iv) any condition requiring a priori anticoagulation, (v) protocol violation.

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 480 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Sayeg-Porto, MD, PhD, Principal Investigator — Hospital dos Servidores do Estado, RJ; Universidade Federal do Rio de Janeiro; Paulo R Benchimol-Barbosa, MD, DSc, Principal Investigator — Universidade Gama Filho; COPPE/UFRJ; Silvia Hoirisch-Clapauch, MD, Principal Investigator — Hospital dos Servidores do Estado, RJ
Locations (1):
- Hospital Federal dos Servidores do Estado, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Hoirisch-Clapauch S, Porto MAS. Early neonatal hypoglycemia prediction according to maternal parameters. Thrombosis Research 131(1): S96, 2013.
- See also: Data presented at the Women's Health Issues in Thrombosis and Hemostasis Meeting, in Vienna, February 2013. — http://www.deepdyve.com/lp/elsevier/p-076-early-neonatal-hypoglycemia-prediction-according-to-maternal-3zQ1tPC9EFct

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment has started in March 2011 at a High-Risk Maternal and Fetal Unit of a tertiary hospital. Enrollment started in May 2011.
Groups:
- Lifestyle Counseling: Daily brisk walking plus a carbohydrate-restricted diet. Patients assigned to the intervention protocol will be instructed to walk briskly for at least 40 minutes seven days a week, to avoid high-carbohydrate meals (such as snacks, candies, fiber-free juices and sugar-sweetened beverages), and to eat at least two daily servings of meat, poultry, fish (e.g. 2 g/kg) or other protein-rich food, starting when they decided to get pregnant and continuing until delivery. Antidepressants will be not discontinued, but patients on paroxetine and sertraline will be switched to fluoxetine.
- Standard Follow-up: Prenatal care will proceed according to the routine. Antidepressants will be not discontinued, but patients on paroxetine and sertraline will be switched to fluoxetine.
Period: Overall Study
Arm/Group | Lifestyle Counseling | Standard Follow-up
Started | 240 | 240
Completed | 159 | 160
Not Completed | 81 | 80
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 0 | 3
Not completed — Multiple pregnancy | 2 | 4
Not completed — Still pregnant when study ended | 13 | 2
Not completed — Did not manage to get pregnant | 64 | 70
Not completed — Had a 2nd trimester loss after accident | 1 | 0

BASELINE CHARACTERISTICS:
Population: Women with recurrent fetal losses in the first trimester
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Counseling | Standard Follow-up | Total
Number analyzed (Participants) | 240 | 240 | 480
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 240 | 240 | 480
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (6) | 33 (8) | 33 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 240 | 240 | 480
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 240 | 240 | 480

OUTCOME MEASURES:

1. Primary Outcome: Neonatal Hypoglycemia
Description: Any glucose level equal or below 40mg/dL at 1, 2 or 4 h after birth, obtained by heelstick.
Time Frame: 1, 2 and 4 h after birth.
Measure: Number; unit: neonates
Units Other Than Participants: blood samples 1, 2 and 4 h after birth
Arm/Group | Lifestyle Counseling | Standard Follow-up
Number analyzed (Participants) | 140 | 91
Number analyzed (blood samples 1, 2 and 4 h after birth) | 420 | 273
neonates | 3 | 15

2. Secondary Outcome: Refractory Hypoglycemia
Description: Any glucose level ≤ 40/dL at 1, 2 or 4 h:
  1. Neonates with hypoglycemia (glucose level equal or below 40 mg/dL at 1, 2 or 4 h) will be offered milk. Neonates unable to suckle, will be treated with intravenous dextrose for one hour.
  2. A new heel stick blood sample will be drawn to assess glucose levels.
  3. Neonates with persistent hypoglycemia will be considered as refractory hypoglycemia.
Time Frame: One hour after feeding or after intravenous dextrose
Population: All hypoglycemic neonates were screened for refractory hypoglycemia. Only neonates born to mothers who were physically inactive and reported excessive carbohydrate consumption displayed refractory hypoglycemia.
Measure: Number; unit: neonates with refractory hypoglycemia
Groups:
- Neonates Born to Mothers Assigned to Protocol Walking+Diet: Neonates with hypoglycemia (blood glucose levels ≤ 40 mg/dL) at 1, 2 or 4 hours after birth
- Neonates Born to Controls: Neonates with hypoglycemia detected 1, 2 or 4 hours after birth
Arm/Group | Neonates Born to Mothers Assigned to Protocol Walking+Diet | Neonates Born to Controls
Number analyzed (Participants) | 3 | 15
neonates with refractory hypoglycemia | 0 | 3

3. Other Pre Specified Outcome: Pregnancy and Neonatal Outcomes
Description: Early miscarriages, 2nd and 3rd trimester losses, preterm deliveries, take-home babies, neonatal hypoglycemia: number of babies
Time Frame: Three years
Measure: Number; unit: participants (babies)
Arm/Group | Lifestyle Counseling | Standard Follow-up
Number analyzed (Participants) | 159 | 160
participants (babies)
  Early Miscarriages | 19 | 62
  Second and Third Trimester Losses | 0 | 7
  Live Born | 140 | 91
  Term | 126 | 57
  Take-home babies | 140 | 83
  Neonatal hypoglycemia | 3 | 15
Statistical Analysis 1: Comparison: Lifestyle Counseling vs Standard Follow-up; Take home babies; Test type: Superiority or Other; p < 0.05, Chi-squared; Odds Ratio (OR) = 3.4, 95% CI 2-sided [1.5 to 7.6], Standard Deviation 1

ADVERSE EVENTS:
Time Frame: From the first prenatal consultation until four hours after delivery. Intervention refers to the mother. The outcome refers to the baby or to the mother.
Groups:
- Standard Follow-up (Mothers); Standard Follow-up (Babies): Prenatal care will proceed according to the routine.
- Lifestyle Counseling (Mothers); Lifestyle Counseling (Babies): Exercise plus a carbohydrate-controlled diet.
Arm/Group | Standard Follow-up (Mothers) | Lifestyle Counseling (Mothers) | Standard Follow-up (Babies) | Lifestyle Counseling (Babies)
Serious Adverse Events (participants affected / at risk) | 36/160 | 10/159 | 84/160 | 22/159
Other Adverse Events (participants affected / at risk) | 0/160 | 0/159 | 0/160 | 0/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Standard Follow-up (Mothers) (N=160) | Lifestyle Counseling (Mothers) (N=159) | Standard Follow-up (Babies) (N=160) | Lifestyle Counseling (Babies) (N=159)
First trimester (Pregnancy, puerperium and perinatal conditions) | 0/0 | 0/0 | 62 | 19 — early miscarriages
Second and third trimester (Pregnancy, puerperium and perinatal conditions) | 0/0 | 0/0 | 7 (7) | 0 — Fetal losses
Gestational diabetes mellitus (Endocrine disorders) | 17 | 3 | 0/0 | 0/0
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 22 | 8 | 0/0 | 0/0
neonatal hypoglycemia (Pregnancy, puerperium and perinatal conditions) | 0/0 | 0/0 | 15/91 | 3/140 — Glucose levels ≤ 40 mg/dL at 1, 2 or 4 hours after birth
neonatal death (Pregnancy, puerperium and perinatal conditions) | 0/0 | 0/0 | 8/91 | 0/140

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No